CLINICAL TRIAL: NCT06517472
Title: Comparison of Pit Picking, Phenol and Combined Pit Picking and Phenol Applications in Pilonidal Sinus Treatment
Status: Recruiting | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Ivstrh 214
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Pilonidal Sinus
Keywords: Pilonidal sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bascom's pit-picking: In the pit-picking technique, midline pits will be excised with minimal tissue removal (skin margin <1 mm). Hairs in the sinuses will be removed along with the curetted tissues. The midline excision areas and secondary pits excised near the midline will be closed with 3-0 polypropylene.
- Crystallized phenol: In crystallized phenol treatment, the pit will be expanded with the help of a clamp, and after confirming it is uncomplicated, hair and infected tissue will be cleaned. Nitrofurazone will be applied to the pit edges. Crystallized phenol will be filled into the sinus with the help of a clamp.
- Combined treatment: In the combined treatment, crystallized phenol will be applied after pit picking, and the pit area will be left to secondary healing.

SUMMARY:
Pilonidal sinus disease is a common condition, and treatment options and outcomes vary greatly. Chronic symptomatic pilonidal sinus disease (PSD) primarily affects young adults and causes work loss. In this study, three treatment methods will be performed: the minimally invasive pit-picking procedure, crystallized phenol application (CPT), and a combined method (minimally invasive pit-picking procedure and CPT). The aim of this study is to compare the effectiveness of these three methods, evaluate short- and long-term results, and determine treatment success, the incidence of postoperative complications, chronic pain levels, recurrence rates, and patient satisfaction. Additionally, the effects of these methods on hospital stay, wound healing time, and workforce loss will also be examined.

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) is common, affecting approximately 26 in 100,000 people. Treatment options and outcomes vary significantly. Chronic symptomatic pilonidal sinus disease primarily affects young adults and leads to substantial work loss. Due to the heterogeneous nature of clinical presentations, finding a single treatment approach for PSD has proven difficult. Future clinical studies might benefit from focusing on the best management strategies rather than the best technique.

Literature indicates that the minimally invasive pit-picking procedure has a general treatment success rate of 68%, with low postoperative complication rates, chronic pain, and high patient satisfaction regarding cosmetic appearance. It is seen as a better option in terms of pain, wound healing time, and complication rates. For simple, uncomplicated pilonidal sinus cases, the pit-picking method is an alternative to flap surgery in terms of wound healing and recurrence.

Particularly for patients with fewer than two pits and no lateral extensions, crystallized phenol application (CPT) is a good alternative to modified Limberg flap surgery and other surgical procedures. CPT, being a minimally invasive procedure performed under local anesthesia, has higher success rates after recurrent applications and shorter hospital stays. Long-term results for CPT treatment are also quite successful. Studies show that in addition to endoscopic pilonidal sinus treatment, crystallized phenol treatment is safe, well-tolerated, and provides quick and lasting recovery without recurrence over the follow-up period.

The presented study aims to compare the effectiveness of three different treatment methods for pilonidal sinus disease: Pit Picking, CPT Application, and Combined Pit Picking and CPT Application. The study will evaluate the short- and long-term results, treatment success, incidence of postoperative complications, chronic pain levels, recurrence rates, and patient satisfaction. Additionally, the study will examine the effects of these methods on hospital stay, wound healing time, and workforce loss. The presented study aims to determine whether minimally invasive procedures and CPT treatment offer better management strategies for pilonidal sinus disease. The findings are expected to contribute to identifying the most suitable treatment method for pilonidal sinus disease.

ELIGIBILITY:
Inclusion Criteria:

* Having two pits or less

Exclusion Criteria:

* With bilateral lateral extension,
* Stage-R with recurrent disease
* Number of pits more than three pits,
* Collagen tissue disease,
* Patients with a postoperative follow-up period of less than 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged 18 and older with pilonidal sinus disease and two or fewer pits, with no previous surgical treatment.
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Success | Up to 12 months post-treatment
  The primary outcome measure will evaluate the effectiveness of three different treatment methods for pilonidal sinus disease: Pit Picking, Crystallized Phenol (CPT) Application, and Combined Pit Picking and CPT Application. Effectiveness will be determined by the absence of disease recurrence and complete healing.
Postoperative Complications | Up to 3 months post-treatment.
  This measure will assess the incidence of postoperative complications such as infection and pain.

SECONDARY OUTCOMES:
Recurrence Rate | Up to 12 months post-treatment
  Evaluation of the rate of disease recurrence after treatment.
Chronic Pain Level | Up to 3 months post-treatment
  Assessment of chronic pain levels in patients following treatment using the Visual Analog Scale (VAS). VAS is a scale from 0 to 10, where 0 represents no pain and 10 represents the worst possible pain. Higher scores indicate worse outcomes.
Patient Satisfaction | Up to 12 months post-treatment
  Measurement of patient satisfaction with the treatment process and outcomes using the Patient and Observer Scar Assessment Scale (POSAS). POSAS is a scale from 1 to 10, where 1 represents the best outcome and 10 represents the worst outcome. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Sehit Prof. Dr. Ilhan Varank Training and Research Hospital, Istanbul, Other, Turkey (Türkiye)